CLINICAL TRIAL: NCT06002906
Title: The Use of Indocyanine Green to Visualize Blood Flow to the Gastrojejunostomy During Bariatric Surgery
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Stryker Endoscopy (Industry)
Responsible Party: Principal Investigator, Allan Okrainec, MD, MHPE, FACS, FRCSC (Principal Investigator), University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-5008
Record Dates: First submitted 2023-08-09; First posted 2023-08-21 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Ulcer, Gastric; Obesity, Morbid
MeSH Terms: conditions — Stomach Ulcer; Obesity, Morbid | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Interventional group (with drug) (Experimental): The interventional group will receive indocyanine green during bariatric surgery inside the operating room before and after making the gastrojejunostomy.
  Interventions: Drug: Indocyanine green; Device: Stryker 1688 AIM system

INTERVENTIONS:
Drug: Indocyanine green — Indocyanine green (ICG) is a safe, sterile, water-soluble molecule that binds to plasma proteins and can be injected intravenously. ICG will be injected intravenously based on the patient's weight prior to and after making the GJ anastomosis and a 10 mL bolus of normal saline will be immediately followed the injection of indocyanine green by an anesthesiologist. A subjective score of 1-5 for perfusion will be assigned by operating surgeons. The RYGB will then be completed by the operating surgeon in their routine fashion.
  Other Names: SPY AGENT GREEN
Device: Stryker 1688 AIM system — The Stryker 1688 AIM system used during laparoscopic surgery which is sensitive in the visible and infrared spectrum. ICG (SPY AGENT™ GREEN) is used with the SPY mode in the Stryker 1688 AIM fluorescence imaging system to perform intraoperative fluorescence angiography.

SUMMARY:
This is an interventional pilot study aimed to evaluate the use of NIF imaging as an intraoperative aid to assess the anastomotic blood flow to the gastric pouch and gastrojejunostomy during Roux-en-Y gastric bypass surgery and to determine its long-term impact on the rate of marginal ulceration, leaks and stricture.

DETAILED DESCRIPTION:
The purpose of this study is to examine intraoperative usefulness of near-infrared light fluorescence imaging with a contrast agent called indocyanine green to improve visualization of blood flow to a surgical connection between the small intestine and stomach (gastrojejunostomy) in patients undergoing gastric bypass surgery. ICG will be given prior to and after making the gastrojejunostomy to examine blood flow and then a subjective perfusion score will be given by the surgeon and assistant during the surgery.

Patients will be recruited before the laparoscopic Roux-en-Y gastric bypass surgery and the study data will be collected prospectively through standard bariatric follow up visits up to 2 years. A mid-term analysis of the procedure and patient outcomes will be performed for quality assurance purposes when half the study patients have undergone intraoperative ICG use. The ICG will be not given if a patient is allergic to sodium iodide or has a history of allergy to iodides because of the risk of a severe allergic reaction.

Participants will be assigned an identifying number to protect confidentiality. Descriptive univariate and multivariate statistical analysis will be performed on all patients satisfying the study's inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to provide informed consent.
* Over the Age of 18.
* Eligible for bariatric surgery in Ontario and deemed an appropriate candidate for RYGB surgery by the bariatric program.
* Commit to follow-up within the bariatric program, including behavioral and dietary modifications designed to aid in sustained weight-loss.
* Treatment of marginal ulcer with the revisional surgery.

Exclusion Criteria:

* Not willing to participate in study
* Contraindication to, or not planned to undergo RYGB
* Known allergy to indocyanine green or Sodium Iodide
* Is participant pregnant or planning to get pregnant in next two years
* Ongoing substance abuse or active smoking
* Bleeding diathesis or Coagulopathy
* Unwilling to take PPI medication Post operatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2027-07-03 (Estimated); Study Completion 2027-07-03 (Estimated)

PRIMARY OUTCOMES:
The applicability of ICG as an indicator of anastomotic blood flow during bariatric surgery. | 2 years
  ICG imaging will be performed intraoperatively using an existing imaging system (1688 Advanced Imaging Modalities (AIM) System (Stryker)), and the images will be assessed by the operating surgeons and as well as by an independent surgeon (part of the study team, independent from the surgery) postoperatively using a subjective assessment of intraoperative Fluorescence Intensity (FI), a 5-point scale to check blood flow of the stomach and small intestine at the new connection. The scale range is 1 to 5 where a score of 1 signifies no fluorescence signal and poor blood supply whereas a score of 5 signifies maximum fluorescence signal and blood supply. Images will also be analyzed postoperatively to obtain an objective score based on fluorescence intensity. The applicability of ICG imaging in the context of RYGB will be assessed based on the inter-observer agreement.

SECONDARY OUTCOMES:
The impact of ICG imaging on the rate of marginal ulcer and other complications (leaks, strictures). | 2 years
  The patients in the Toronto Western Hospital as per the standard care of bariatric program will be followed for up to 2 years following surgery to identify any complications including marginal ulcerations. Data is collected prospectively at the study site. The investigator will also use the data from the 5-point scale scoring system reference above to determine the correlation between the scores and the occurrence of marginal ulcers and any other complications (leaks, strictures).
To evaluate the safety of routine use of NIF imaging using ICG in bariatric patients. | 30 days
  Based on the literature, the investigator does not anticipate intra-operative or injection-related adverse effects. Nevertheless, the investigator will use the existing database that collects postoperative outcomes for 30 days to identify adverse events, if any.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Okrainec, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No